CLINICAL TRIAL: NCT05824078
Title: Outcomes of Perilunate Injury Management: Open vs Arthroscopic Approach
Brief Title: Perilunate Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nicole Zelenski, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005088
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Perilunate Injury
Keywords: Carpus; Arthroscopy; Open surgery
MeSH Terms: interventions — Arthroscopy; Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open procedure (Active Comparator): The study intervention involved in this project is the randomized allocation of the patient who requires surgical treatment of their perilunate injury to receive either an open or arthroscopic approach for the procedure.
  Once the patient is in agreement to have surgery and has consented to partake in the study, they will be randomly allocated to either open perilunate surgery or arthroscopic perilunate surgery.
  Both surgical approaches are well-recognized, common, standard-of-care procedures.
  Interventions: Procedure: Open Surgery
- Arthroscopic Procedure (Active Comparator): The study intervention involved in this project is the randomized allocation of the patient who requires surgical treatment of their perilunate injury to receive either an open or arthroscopic approach for the procedure.
  Once the patient is in agreement to have surgery and has consented to partake in the study, they will be randomly allocated to either open perilunate surgery or arthroscopic perilunate surgery.
  Both surgical approaches are well-recognized, common, standard-of-care procedures.
  Interventions: Procedure: Arthroscopic surgery

INTERVENTIONS:
Procedure: Arthroscopic surgery — Arthroscopic approach involves smaller incision, offering less traumatic procedures and faster healing, but due to the limited space in this closed field with significant vasculature and nerve distribution, scoping has increased risk for iatrogenic injuries.
  Arms: Arthroscopic Procedure
Procedure: Open Surgery — The open approach requires dissection of capsuloligamentous structures, which can lead to stiffness of the joint due to capsular scarring as it heals. However, it offers good visual field when treating the injury, allowing maneuverability to avoid iatrogenic soft tissue injuries.
  Arms: Open procedure

SUMMARY:
Perilunate injuries can be debilitating injuries that involve the carpus. These can limit patients' functionality both acutely and long-term. Not only do their potential for nerve injury increase risk of lasting weakness and chronic pain, but their complex surrounding involving the carpus also leads to potential for misalignment when healing. The approach for treating perilunate injuries often relies on internal fixation, prompting the need for surgery. However, there is no clear recommendation for whether to pursue open or arthroscopic surgery as both offer benefits and pose risks.

The aim of this study is to determine the similarities and differences in outcomes for management of perilunate injuries.

DETAILED DESCRIPTION:
Perilunate injuries are those that affect the wrist, which can be debilitating to patients. Often, these injuries require surgical treatment, which can either be performed open or arthroscopic. There is currently no consensus for which approach offers better outcomes. Therefore, this study will allocate patients who require surgical treatment of perilunate injuries to either open or arthroscopic surgical intervention to compare their outcomes. The results will offer insight into the compromises made with each surgical approach and create a foundation orthopedic surgeons can leverage to decide how to manage a patient to ensure best possible outcomes.

This study will involve 12 patients who were identified as having perilunate injuries requiring orthopedic surgical treatment. Their participation will involve consenting to be randomly allocated to the surgical approach, and they will be asked to complete commonly used orthopedic surveys (eg DASH score) that are used to evaluate the functional healing of their injury. They will be followed for up to 1 year after their surgery. A chart review will be conducted to follow their progress and surgical outcomes.

Patients will be recruited from Grady Memorial Hospital. No specimens will be collected or banked for this study.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years old and older).
* Patients requiring surgical intervention for a perilunate injury will be consented and then randomly allocated to either open or arthroscopic surgery.

Exclusion Criteria:

* Prisoners will not be included in this study.
* Patients younger than 18 years old and pregnant patients will be excluded from this review.
* Patients who require specific surgical approach for their treatment, cannot be randomly allocated to one of the study arms, so will be excluded from this study.
* The study will not include data from minors, cognitively impaired individuals, or individuals who are vulnerable to coercion or under influence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Pain Numeric Rating Scale (NRS) | 12 weeks post-operation
  The numeric rating scale is one of the most commonly used pain scales in medicine. The NRS consists of a numeric version of the visual analog scale. The most common form of the NRS is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible.

SECONDARY OUTCOMES:
Range of motion | 12 weeks post-operation
  Range of motion (ROM) means the extent or limit to which a part of the body can be moved around a joint or a fixed point; the totality of movement a joint is capable of doing. A range of motion test, also called a flexibility test, is used to measure the degree of movement of a joint. A goniometer is an instrument that is used to measure the range of motion of a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Zelenski, MD, Principal Investigator — Assistant Professor; Eric R Wagner, MD, Principal Investigator — Assistant Professor
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No